CLINICAL TRIAL: NCT05747560
Title: Study on the Effect of Dietary Supplements on Height Improvement in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Fengqin Feng, Professor Feng, Zhejiang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Feng8898
Record Dates: First submitted 2023-02-04; First posted 2023-02-28 (Actual); Last update posted 2023-03-07 (Actual); Status verified 2023-03

CONDITIONS: Body Height; Child, Only
MeSH Terms: interventions — Huang Qi

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Participants in the Placebo will consume buckwheat at a dose of 500 mg, twice a day (morning and evening) for 6 months.
  Interventions: Dietary Supplement: Buckwheat
- Astragalus extract (Active Comparator): Participants in the Astragalus extract will take dietary supplement with astragalus extract at a dose of 450 mg, twice a day for the same duration.
  Interventions: Dietary Supplement: Astragalus extract
- Wolfiporia extract (Experimental): Participants in the Wolfiporia extract will take dietary supplement with wolfiporia extract at a dose of 15 g, twice a day for the same duration.
  Interventions: Dietary Supplement: Wolfiporia extract

INTERVENTIONS:
Dietary Supplement: Buckwheat — Take buckwheat at a dose of 500 mg twice a day for 6 months.
  Arms: Placebo
Dietary Supplement: Astragalus extract — Take astragalus extract at a dose of 450 mg twice a day for 6 months.
  Arms: Astragalus extract
Dietary Supplement: Wolfiporia extract — Take wolfiporia extract product at a dose of 15 g twice a day for 6 months.
  Arms: Wolfiporia extract

SUMMARY:
With the increasing improvement of living standard, more and more people are concerned about the body height of their children. It has been reported that 542 out of 1000 children (54.2%) failed to meet the standards of height. Moreover, nearly 80% was disappointed with the height of their children. The body height of child is mainly influenced by 60% of genetic factors (6 out of 10) and 40% of acquired factors which includes nutrition, exercise, sleep, psychology, disease and so on. Therefore, it is an important way to solve the problem by regulating the acquired factors. At present, inject growth hormone (GH) for children is the main way to solve the problem of children's body weight. However, high price, complex operation skills, and side effects limits the implication of GH. Additionally, the effect of traditional Chinese medicine therapy, exercise therapy, and dietary supplement are of dubious benefit and without clinical support. Elevated insulin like growth factor-1 (IGF-1) levels in the human body have been recognized as one of the core criteria for evaluating body enhancement therapy. Currently, there is no dietary supplement intervention to enhance the sensitivity of GH receptor and IGF-1 receptor. The goal of this clinical trial is to test the effect of dietary supplements on height improvement in children (aged 8-15 years of both genders). The main question it aims to answer is: Study the effect of dietary supplements (a formula based on enhancing the sensitivity of GH receptor and IGF-1 receptor) on height improvement in children by.

Participants will be randomly divided into three groups: Placebo, Astragalus extract, and Wolfiporia extract.

1. Participants in the Placebo will consume placebo (a look-alike substances that contains no active drug) at a dose of 500 mg, twice a day (morning and evening) for 6 months. Participants in the Astragalus extract will take dietary supplement with astragalus extract at a dose of 450 mg, twice a day for the same duration. Participants in the Wolfiporia extract will take dietary supplement with wolfiporia extract at a dose of 15 g, twice a day for the same duration.
2. Taken blood sample at the timepoint of baseline (Day 0), intermediate point (Day 90), intervention end point (Day 180)) to detect biochemical markers, as well as body height and weight, and skeletal age.
3. Throughout the trial, subjects were asked to keep their usual lifestyle, food, and physical exercise and not took any dietary supplements.

Researchers will compare the effects of Placebo with Astragalus extract, placebo with Wolfiporia extract, and Astragalus extract with Wolfiporia extract to see if Astragalus extract and Wolfiporia extract increase children's height, and whether Astragalus extract or Wolfiporia extract is more works well.

ELIGIBILITY:
Inclusion Criteria:

1. Body height: from the 10th to the 75th;
2. Skeletal age: bone age and actual age ±1.

Exclusion Criteria:

1. Treated with growth hormone;
2. Sexual precocity;
3. Abnormal liver and kidney function;
4. IGF levels: below -2SD and above +2SD;
5. IGF BP3 level: below -2SD;
6. Growth hormone deficiency;
7. Diagnosed genetic disease;
8. BMI: Underweight or obese;
9. Abnormal thyroid function.

Ages: 8 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 90 (Estimated)
Dates: Start 2023-06-20 (Estimated); Primary Completion 2023-12-20 (Estimated); Study Completion 2023-12-30 (Estimated)

PRIMARY OUTCOMES:
Change from baseline body height at 6 months | Baseline (Day 0), Intervention end point (Day 180)
  Determination of the change of body height of the participants at 6 months.

SECONDARY OUTCOMES:
Change from baseline skeletal age at 6 months | Baseline (Day 0), Intervention end point (Day 180)
  Determination of the change of skeletal age of the participants at 6 months.
Change from baseline body weight at 6 months | Baseline (Day 0), Intervention end point (Day 180)
  Determination of the change of body weight of the participants at 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Fengqin Feng, Study Chair — Zhejiang University
Locations (1):
- College of Biosystems Engineering and Food Science, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Undecided